CLINICAL TRIAL: NCT06393140
Title: The Study on the Mechanism of Radiotherapy-elicited Immune Response
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, professor, Fudan University
Other Study IDs: ESO-shanghai 23
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Carcinoma Salivary Gland Type; Radiotherapy
Keywords: Esophageal Carcinoma; Tumor-draining lymph nodes; Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Histological specimens of tumors derived from surgical or metastatic sites
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy plays an important role in multidisciplinary treatment of esophageal cancer. Data from many laboratories indicate that local radiation produces systemic, immune-mediated anti¬tumour and, potentially, antimetastatic effects. Additionally, the combination of local radiotherapy and immune-modulation can augment local tumour control and cause distant (abscopal) antitumour effects through increased tumour-antigen release and antigen-presenting cell (APC) cross-presentation, improved dendritic-cell (DC) function, and enhanced T cell priming. The generation of an effective antitumor immune response requires the presentation of tumor antigens to naïve CD8+ cells in tumor-draining lymph nodes (TDLN) . Tumor-draining lymph nodes, however, are often subject to the immunosuppressive activity of tumor-derived factors, such as cytokines and other bioactive molecules from tumor cells and their associated leukocytes in the primary tumor site that contribute to the overriding of effective rejection mechanisms. Thus, in TDLN a T cell tolerance rather than a T cell activation often occurs, thereby preventing immune attack and facilitating local tumor progression.

DETAILED DESCRIPTION:
In this study, the investigators collect clinical and biological evidence to interpret the impact of radiotherapy on tumor regression and immunity, and identify key molecular features and immune landscape patterns to characterize patients sensitive/resistant to radiotherapy; and define the dynamic changes occurring in TME and lymph node after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. new diagnosis locoregional esophageal cancer;
2. pathologic diagnosis is squamous carcinoma;
3. Patients had received either neoadjuvant or definitive radiotherapy
4. tumor and lymph node tissue can be collected and can be conducted with single cell RNA (scRNA)-sequencing and other sequencings.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Unable or rejection to receive radiotherapy or unable to comply with study requirements or follow-up schedule.
3. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Genetic signature of patients who had received neoadjuvant or definitive radiation therapy | 4-year
  Detailed mechanism of radiation-activated immunity under single-cell sequencing.gene mutations, copy number variants.

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, MD, Study Director — Fudan University
Locations (1):
- Fudan University Shanghai cancer center, Shanghai, China